CLINICAL TRIAL: NCT07344233
Title: Brain-to-brain Neurofeedback During Naturalistic Dynamic Stimuli to Reduce Craving in Heroin Addiction
Brief Title: Neurofeedback During Naturalistic Stimuli to Reduce Craving in Heroin Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rita Goldstein, Professor of Psychiatry and Neuroscience, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: GCO 22-1694; R21DA058801 (NIH)
Record Dates: First submitted 2026-01-14; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Substance Use Disorder; Heroin Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real Neurofeedback (Experimental): Participants receive real-time fMRI neurofeedback reflecting their own brain activity during a drug-related movie.
  Interventions: Behavioral: Real-time fMRI Neurofeedback
- Sham (yolked) Neurofeedback (Sham Comparator): Participants receive sham real-time fMRI neurofeedback yoked to a matched participant and unrelated to their own brain activity.
  Interventions: Behavioral: Sham Real-time fMRI Neurofeedback

INTERVENTIONS:
Behavioral: Real-time fMRI Neurofeedback — Real-time feedback reflecting the similarity between participant's brain activity patterns and a predefined target while viewing a drug-related movie.
  Arms: Real Neurofeedback
Behavioral: Sham Real-time fMRI Neurofeedback — Real-time feedback yoked to another participant and not reflective of the participant's own brain activity.
  Arms: Sham (yolked) Neurofeedback

SUMMARY:
Support groups are an important component of addiction treatment, where individuals at more stable stages of their recovery help others by sharing personal experiences. This phenomenon suggests that the brain states of individuals further along in their recovery process may be useful in guiding those who are at an earlier stage. In this project, the researchers will test this idea and develop a personalized therapeutic tool based on real-time fMRI neurofeedback, whereby individuals with heroin use disorder (iHUD) early in treatment will learn to modulate their own brain state to more closely align with iHUD who are at later stages of treatment. Specifically, iHUD exhibit heightened reactivity to naturalistic drug cues in brain networks underlying salience attribution, reward processing, executive function and others. This fMRI brain hyperactivity pattern is reduced, concomitant with craving reductions, with about 3 months of inpatient treatment. In this neurofeedback project, iHUD who are beginning treatment will view naturalistic drug cues and receive feedback about how similar their brain activity is to the target recovery pattern, learning to modulate their own brain activity to reduce drug cue reactivity and craving. This study will offer insights into the mechanisms of recovery in addiction, particularly as coordinated across individuals with shared experience and goals. If successful, the neurofeedback-based training may lead to new brain-based and personalized tools for recovery in this devastating disorder.

ELIGIBILITY:
Inclusion criteria:

* Ability to understand, give informed consent and perform the tasks
* males and females 18-64 years of age at the time of enrollment in the study
* DSM-5 diagnosis of opioid use disorder with heroin as the primary drug of choice
* currently enrolled in a treatment facility for heroin use as the primary concern
* 2-4 week abstinence from non-prescribed opioid use/stabilized on medication assisted therapy (MAT) using either methadone and/or buprenorphine.

Exclusion criteria:

* present or past history of a neurodevelopmental, neurological, or a psychotic disorder
* head trauma with loss of consciousness for more than 30 min
* use of medications (current or in the last 6 months) with known CNS effects which may alter cerebral function, with the exception of psychotropics for the treatment of pain/depression/anxiety/PTSD (e.g. SSRIs) or as otherwise determined by the Principle Investigator
* current medical illness and/or evident infection
* being pregnant or nursing
* contraindications to the MRI environment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Cue/movie-induced craving score | Immediately before and immediately after neurofeedback procedure
  Self-reported ratings of heroin craving on a 0-9 point scale, with higher scores indicating higher craving.

SECONDARY OUTCOMES:
Neurofeedback Score Change | During each 20 minute neurofeedback training session. Participants complete 8 neurofeedback sessions over the course of 4 consecutive days.
  Change in neurofeedback performance, reflecting participants' ability to modulate brain activity toward the predefined target pattern. Neurofeedback scores range 0-100, with higher scores indicating more similar brain activity to the target pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Goldstein, PhD, Principal Investigator — NARC@mssm.edu
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Specify Other Mechanism Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to NARC@mssm.edu. To gain access, data requestors will need to sign a data access agreement.